CLINICAL TRIAL: NCT01670825
Title: Randomized, Double-blind, Comparative-effectiveness Study Comparing Corticosteroid Injections to Pulsed Radiofrequency for Occipital Neuralgia
Brief Title: Pulsed Radiofrequency vs. Steroid Injections for Occipital Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven P. Cohen, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 373481-3
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Occipital Neuralgia
Keywords: Occipital neuralgia; corticosteroid injection; pulsed radiofrequency
MeSH Terms: interventions — Pulsed Radiofrequency Treatment; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed radiofrequency + local anesthetic injection (Experimental): Local anesthetic injection plus pulsed radiofrequency over each affected occipital nerve
  Interventions: Procedure: Pulsed radiofrequency; Drug: Local anethestic injection
- Corticosteroid injection + sham pulsed radiofrequency (Active Comparator): Injection with corticosteroid and local anesthetic over the occipital nerve(s)plus "sham" pulsed radiofrequency
  Interventions: Drug: Corticosteroid injection; Drug: Local anethestic injection

INTERVENTIONS:
Procedure: Pulsed radiofrequency — Local anesthetic injection and pulsed radiofrequency treatment x 6 minutes over each affected occipital nerve
  Arms: Pulsed radiofrequency + local anesthetic injection
Drug: Corticosteroid injection — Corticosteroid and local anesthetic injection plus sham pulsed radiofrequency over each affected occipital nerve
  Arms: Corticosteroid injection + sham pulsed radiofrequency
Drug: Local anethestic injection
  Other Names: Local anethestic injection that both arms will receive

SUMMARY:
The aim of this study is to determine whether pulsed radiofrequency or steroids are better for occipital neuralgia. Seventy-six patients with ON or migraine with tenderness over the occipital nerve who respond to occipital nerve blocks (hereafter included under the broad category "ON") will be randomized in a 1:1 ratio to receive either corticosteroid and local anesthetic injections (n=38) or local anesthetic and PRF of the occipital nerve(s) (n=38) for occipital neuralgia. Both patients and the treating & evaluating physicians will be blinded. The first follow-up visit will be at 6 weeks. Patients who obtain significant pain relief will remain in the study. Those patients who fail to obtain any benefit will exit the study and be allowed to crossover to the other treatments or receive alternative care. The second follow-up will be at 3 months and the final follow-up will be at 6-months post-procedure.

DETAILED DESCRIPTION:
Up to 76 patients referred to one of the participating pain clinic with occipital neuralgia, or migraines with occipital nerve tenderness (dual diagnoses) will be randomized in a 1:1 ratio by a computer generated randomization table to receive one of two treatments. Treatments will be randomized at each institution. Within each group, those patients with plain occipital neuralgia, and those with occipital neuralgia with migraines, will be sub-randomized in the same 1:1 ratio. Diagnosis of ON will be made by low-volume (< 3 mL bupivacaine per nerve). Our criterion for a positive response will be > 50% pain relief lasting at least 3 hours. Those individuals who have symptoms in the distribution of both the greater and lesser occipital nerves will receive treatment of both nerves. The greater occipital nerve is more frequently affected than the lesser nerve.

Half (n=38) of the patients will be allocated to receive local anesthetic & corticosteroid injections at each nerve (group I), with an equal number allocated to receive local anesthetic & PRF at each (group II). In those patients who request sedation, an intravenous will be inserted and light sedation administered with low doses of midazolam and fentanyl, in accordance with our standard clinic practice. Treatment in all patients will be accomplished using 20-gauge radiofrequency needles with 10 mm active tips. Prior to treating, electrical stimulation will be performed to ensure ample proximity to the targeted nerve(s), with our target threshold being concordant stimulation at < 0.3 volts at each site.

Once proper needle position is ensured, those in group I will receive an injection at each nerve containing 30 mg of depomethylprednisolone mixed with 2 mL of a 50:50 mixture of 2% lidocaine and 0.5% bupivacaine (2.75 mL). Anywhere between 1 and 4 nerves can be injected, with 4 nerves being targeted if a patient had bilateral lesser and greater occipital nerve involvement. This will be followed by 3 cycles of sham PRF at 120 s per cycle, with slight (approximately 30o electrode adjustments between cycles. For sham PRF, no electrical field or heat is generated (i.e. the machine is not set to any radiofrequency cycle after stimulation), but the cycle times (120 s per cycle) are adhered to (i.e. we will wait a total of 6", 2" per cycle). Those patients in group II will receive injections at each nerve containing 2.75 mL of a solution with 2 mL of 50:50 2% lidocaine and 0.5% bupivacaine + 0.75 mL saline (2.75 mL), followed by 3 cycles of PRF using the following standard settings: voltage output 40-60 V; 2 Hz frequency; 20 ms pulses in a 1-second cycle, 120 second duration per cycle; impedance range between 150 and 400 Ohms; and 42o C plateau temperature.

No patient will be prescribed additional medications or therapy between their procedure and first follow-up. However, they will be allowed to remain on their current, stable analgesic regimen. Rescue medications will consist of tramadol 50 mg 1 to 2 tablets every 6 hours PRN (up to 8/d) and/or acetaminophen or a non-steroidal anti-inflammatory drug such as ibuprofen, diclofenac or ketorolac on an "as needed" basis.

Follow-ups will be performed by a physician blinded to treatment allocation. A preliminary follow-up will be performed at weeks. The first full follow-up visit will be scheduled 6-weeks from the start of treatment. A positive outcome will be defined as a > 50% decrease in headache coupled with a positive satisfaction rating (> 3 on a 0-5 scale). Subjects who obtain a positive outcome at their initial 6-week follow-up visit will remain in the study and return for their 3-month follow-up visit. Those with a negative outcome will exit the study "per protocol" to receive standard care. Subjects who obtain a positive outcome at 1-month but experience a recurrence before their 3-month follow-up visit will also exit the study per protocol, with their final outcome measures recorded before they receive standard care. Those who obtain a positive outcome at 3-months will remain in the study for their final 6-month follow-up, while those who obtain a negative outcome will exit the study. Unblinding for both patients and the treating physician will be after the patient exits the study or after their final follow-up visit for those with continued benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years
2. Occipital neuralgia diagnosed based on history & physical exam and diagnostic local anesthetic blocks, or migraine with occipital nerve(s) tenderness that responds to diagnostic blocks.

   a. Greater or equal to 50% relief based on diagnostic local anesthetic block of the greater and/ or lesser occipital nerves that lasts for at least 90 minutes with lidocaine or 3 hours with bupivacaine or ropivacaine 20
3. Baseline Numerical Rating Scale average pain score > 4/10
4. Frequency of greater or equal to 4/10 pain for at least 10 days per month

Exclusion Criteria:

1. Untreated coagulopathy
2. Automatic implantable cardiac defibrillator or pacemaker that cannot be temporarily disabled for medical reasons
3. Previous pulsed radiofrequency
4. Other sources of headache, such as tension-type headache, cervicogenic headache, migraine headache without occipital neuralgia, and other causes (e.g. tumors, congenital abnormalities etc.). Those that can be confused with ON must be excluded based on history and exam (e.g. cervicogenic headaches), symptoms (tension-type headache), response to blocks (all of the above); and lab work (temporal arteritis, which would be confirmed by biopsy after an elevated erythrocyte sedimentation rate).
5. Serious medical or uncontrolled or severe psychiatric -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

REFERENCES:
- [Background] Huang JH, Galvagno SM Jr, Hameed M, Wilkinson I, Erdek MA, Patel A, Buckenmaier C 3rd, Rosenberg J, Cohen SP. Occipital nerve pulsed radiofrequency treatment: a multi-center study evaluating predictors of outcome. Pain Med. 2012 Apr;13(4):489-97. doi: 10.1111/j.1526-4637.2012.01348.x. Epub 2012 Mar 5. PMID 22390409
- [Background] Vanelderen P, Rouwette T, De Vooght P, Puylaert M, Heylen R, Vissers K, Van Zundert J. Pulsed radiofrequency for the treatment of occipital neuralgia: a prospective study with 6 months of follow-up. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):148-51. doi: 10.1097/aap.0b013e3181d24713. PMID 20301822
- [Background] Choi HJ, Oh IH, Choi SK, Lim YJ. Clinical outcomes of pulsed radiofrequency neuromodulation for the treatment of occipital neuralgia. J Korean Neurosurg Soc. 2012 May;51(5):281-5. doi: 10.3340/jkns.2012.51.5.281. Epub 2012 May 31. PMID 22792425
- [Derived] Cohen SP, Peterlin BL, Fulton L, Neely ET, Kurihara C, Gupta A, Mali J, Fu DC, Jacobs MB, Plunkett AR, Verdun AJ, Stojanovic MP, Hanling S, Constantinescu O, White RL, McLean BC, Pasquina PF, Zhao Z. Randomized, double-blind, comparative-effectiveness study comparing pulsed radiofrequency to steroid injections for occipital neuralgia or migraine with occipital nerve tenderness. Pain. 2015 Dec;156(12):2585-2594. doi: 10.1097/j.pain.0000000000000373. PMID 26447705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Started | 42 | 39
Completed | 42 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (10.72) | 41.08 (13.61) | 41.37 (12.16)
Gender [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 41 | 38 | 79
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Occipital Pain 6 Weeks After the Start of Treatment
Description: The change in the numeric pain scale score from baseline to 6 weeks after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 42 | 39
units on a scale | 3.068 (2.431) | 3.738 (2.415)

2. Primary Outcome: Change in Worst Occipital Pain 6 Weeks After the Start of Treatment
Description: as for outcome 1
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pulsed Radiofrequency + Local Anesthetic Injection: Local anesthetic injection plus pulsed radiofrequency over each affected occipital nerve
  Pulsed radiofrequency: Local anesthetic injection and pulsed radiofrequency treatment x 6 minutes over each affected occipital nerve
  Local anethestic injection
- Corticosteroid Injection + Sham Pulsed Radiofrequency: Injection with corticosteroid and local anesthetic over the occipital nerve(s)plus "sham" pulsed radiofrequency
  Corticosteroid injection: Corticosteroid and local anesthetic injection plus sham pulsed radiofrequency over each affected occipital nerve
  Local anethestic injection
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 41 | 39
units on a scale | 5.354 (3.165) | 6.064 (3.226)

3. Primary Outcome: Change in Average Occipital Pain 6 Months After the Start of Treatment
Description: The change in the numeric pain scale score from baseline to 6 months after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 42 | 39
units on a scale | 4.312 (2.232) | 4.765 (1.998)

4. Primary Outcome: Change in Worst Occipital Pain 6 Months After the Start of Treatment
Description: This outcome measures the change in the numeric pain scale score from baseline to 6 months after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 42 | 39
units on a scale | 6.705 (2.892) | 7.541 (2.416)

5. Primary Outcome: Change in Average Occipital Pain 3 Months After the Start of Treatment
Description: This outcome measures the change in the numeric pain scale score from baseline to 3 months after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 40 | 37
units on a scale | 3.791 (2.573) | 4.441 (2.237)

6. Primary Outcome: Change in Worst Occipital Pain 3 Months After the Start of Treatment
Description: as for outcome 5
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 40 | 37
units on a scale | 5.850 (3.292) | 7.149 (2.967)

7. Primary Outcome: Change in Average Occipital Pain 2 Weeks After the Start of Treatment
Description: This outcome measures the change in the numeric pain scale score from baseline to 2 weeks after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 2 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 42 | 39
units on a scale | 2.495 (2.094) | 3.694 (2.221)

8. Primary Outcome: Change in Worst Occipital Pain 2 Weeks After the Start of Treatment
Description: as for outcome 7
Time Frame: From baseline to 2 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 42 | 39
units on a scale | 4.726 (2.528) | 5.846 (2.618)

9. Primary Outcome: Change in Overall Average Headache Pain 2 Weeks After the Start of Treatment
Description: as for outcome 7
Time Frame: From baseline to 2 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 25 | 20
units on a scale | 3.392 (2.106) | 4.220 (2.496)

10. Primary Outcome: Change in Overall Worst Headache Pain 2 Weeks After the Start of Treatment
Description: as for outcome 7
Time Frame: From baseline to 2 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 25 | 20
units on a scale | 5.540 (2.669) | 6.650 (2.744)

11. Primary Outcome: Change in Overall Average Headache Pain 6 Weeks After the Start of Treatment
Description: This outcome measures the change in the numeric pain scale score from baseline to 6 weeks after treatment. The scale ranges from 0-10. The minimum score is 0 which is defined as no pain and the maximum score is 10, which is defined as the worst pain imaginable. The best possible outcome would be a 0. The worst possible outcome would be a 10.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 20
units on a scale | 3.678 (2.448) | 4.410 (2.544)

12. Primary Outcome: Change in Overall Worst Overall Headache Pain 6 Weeks After the Start of Treatment
Description: as for outcome 11
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 20
units on a scale | 6.583 (3.202) | 6.825 (3.109)

13. Primary Outcome: Change in Overall Average Headache Pain 3 Months After the Start of Treatment
Description: as for outcome 5
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 18
units on a scale | 4.000 (2.870) | 4.694 (2.480)

14. Primary Outcome: Change in Overall Worst Headache Pain 3 Months After the Start of Treatment
Description: as for outcome 5
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 18
units on a scale | 6.522 (3.232) | 7.417 (2.952)

15. Primary Outcome: Change in Overall Average Headache Pain 6 Months After the Start of Treatment
Description: as for outcome 4
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 18
units on a scale | 6.761 (3.096) | 7.556 (2.623)

16. Primary Outcome: Change in Overall Worst Headache Pain 6 Months After the Start of Treatment
Description: as for outcome 4
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 18
units on a scale | 6.761 (3.096) | 7.556 (2.623)

17. Secondary Outcome: Change in the Presence of Insomnia 6 Weeks After the Start of Treatment Measured Using the Athens Insomnia Scale.
Description: This outcome will measure the participant's perceived improvement in sleep using the Athens Insomnia Scale. Scores in this scale can range from 0 to 24. 0 being the best possible outcome and 24 being the worst possible outcome. A score greater than or equal to 6 indicates a presence of insomnia.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 40 | 38
units on a scale | 10.025 (5.972) | 8.132 (5.297)

18. Secondary Outcome: Change in the Presence of Insomnia 3 Months After the Start of Treatment Measured Using the Athens Insomnia Scale.
Description: as for outcome 17
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 9.539 (6.043) | 9.069 (5.955)

19. Secondary Outcome: Change in the Presence of Insomnia 6 Months After the Start of Treatment Measured Using the Athens Insomnia Scale.
Description: as for outcome 17
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 9.256 (6.210) | 9.431 (5.765)

20. Secondary Outcome: Change in the Severity of Depression 6 Weeks After the Start of Treatment Measured Using the Beck's Depression Inventory
Description: This outcome will measure the change in severity of depression using the Beck's Depression Inventory. Scores in this inventory can range from 0 to 63. 0 being the best possible outcome and 63 being the worst possible outcome. A score between 14 and 19 indicates mild depression and a score greater than or equal 29 indicates severe depression.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 40 | 38
units on a scale | 12.775 (11.079) | 10.842 (9.945)

21. Secondary Outcome: Change in the Severity of Depression 3 Months After the Start of Treatment Measured Using the Beck's Depression Inventory
Description: as for outcome 20
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 11.333 (10.207) | 11.972 (10.287)

22. Secondary Outcome: Change in the Severity of Depression 6 Months After the Start of Treatment Measured Using the Beck's Depression Inventory
Description: as for outcome 20
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 12.590 (10.684) | 12.250 (10.103)

23. Secondary Outcome: Severe Headache Frequency for Migraine Headaches 6 Weeks After the Start of Treatment Measured Asking the Number of Severe Headaches in the Past Week.
Description: This outcome will measure the number of days the patient has severe migraine headaches in the week (7 days) prior to the 6 week follow-up visit. A severe headache is defined as a headache with a score greater than or equal to 7 on the numeric pain scale.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 24 | 20
days | 1.708 (1.958) | 1.810 (2.421)

24. Secondary Outcome: Severe Headache Frequency for Occipital Neuralgia Headaches 6 Weeks After the Start of Treatment Measured Asking the Number of Severe Headache Days 1 Week Prior to Study Visit
Description: This outcome will measure the number of days the patient has severe occipital neuralgia headaches in the week (7 days) prior to the 6 week follow-up visit. A severe headache is defined as a headache with a score greater than or equal to 7 on the numeric pain scale.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 41 | 38
days | 1.436 (2.237) | 1.436 (2.087)

25. Secondary Outcome: Severe Headache Frequency for Migraine Headaches 3 Months After the Start of Treatment Measured Asking the Number of Severe Headache Days 1 Week Prior to Study Visit
Description: This outcome will measure the number of days the patient has severe migraine headaches in the week (7 days) prior to the 3 month follow-up visit. A severe headache is defined as a headache with a score greater than or equal to 7 on the numeric pain scale.
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 23 | 19
days | 2.087 (2.109) | 2.263 (2.232)

26. Secondary Outcome: Severe Headache Frequency for Occipital Neuralgia Headaches 3 Months After the Start of Treatment Measured Asking the Number of Severe Headache Days 1 Week Prior to Study Visit
Description: as for outcome 24
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 37
days | 1.846 (2.335) | 1.919 (2.046)

27. Secondary Outcome: Severe Headache Frequency for Migraine Headaches 6 Months After the Start of Treatment Measured Asking the Number of Severe Headache Days 1 Week Prior to Study Visit
Description: This outcome will measure the number of days the patient has severe migraine headaches in the week (7 days) prior to the 6 month follow-up visit. A severe headache is defined as a headache with a score greater than or equal to 7 on the numeric pain scale.
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 23 | 19
days | 2.044 (2.099) | 2.368 (2.409)

28. Secondary Outcome: Severe Headache Frequency for Occipital Neuralgia Headaches 6 Months After the Start of Treatment Measured Asking the Number of Severe Headache Days 1 Week Prior to Study Visit
Description: as for outcome 24
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 37
days | 2.128 (2.308) | 2.162 (2.154)

29. Secondary Outcome: Disability Due to Headaches 6 Weeks After the Start of Treatment Measured Using the Headache Impact Scale
Description: This outcome measures what the patient feels they cannot do because headaches. This outcome is measured using the Headache Impact Test. Scores in this test range from range from 36 to 78, with higher scores indicating greater negative impact. A score of less than 50 indicates minimal impact, while a score greater than or equal to 60 indicates headaches are severely impacting one's life.
Time Frame: From baseline to 6 weeks after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 40 | 38
units on a scale | 60.087 (7.972) | 59.553 (9.093)

30. Secondary Outcome: Disability Due to Headaches 3 Months After the Start of Treatment Measured Using the Headache Impact Scale
Description: as for outcome 29
Time Frame: From baseline to 3 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 59.718 (9.761) | 60.556 (10.814)

31. Secondary Outcome: Disability Due to Headaches 6 Months After the Start of Treatment Measured Using the Headache Impact Scale
Description: as for outcome 29
Time Frame: From baseline to 6 months after the start of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Number analyzed (Participants) | 39 | 36
units on a scale | 59.641 (10.251) | 61.389 (8.800)

ADVERSE EVENTS:
Arm/Group | Pulsed Radiofrequency + Local Anesthetic Injection | Corticosteroid Injection + Sham Pulsed Radiofrequency
Serious Adverse Events (participants affected / at risk) | 3/42 | 6/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Radiofrequency + Local Anesthetic Injection (N=42) | Corticosteroid Injection + Sham Pulsed Radiofrequency (N=39)
Dizzines (Nervous system disorders) | 0 (0) | 1 (1) — 1 person in the steroid group experienced dizziness after the procedure.
Swelling at injection site (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — 2 people in the steroid group had swelling at the injection site
Worsening of headached (Nervous system disorders) | 1 (1) | 2 (2) — 2 people in the steroid group and 1 in the PRF group experienced worsening of headache after procedure.
Vomiting/blurred vision (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes